CLINICAL TRIAL: NCT03662477
Title: Effect of Autologous NK Cell Immunotherapy on Advanced Lung Adenocarcinoma With EGFR Mutation: a Preliminary Clinical Study
Brief Title: Effect of NK Cell Immunotherapy on Advanced Lung Adenocarcinoma Adenocarcinoma With EGFR Mutation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Fifth People's Hospital (Other)
Responsible Party: Principal Investigator, LiuTao, Principal Investigator, Shenzhen Fifth People's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Shenzhen Fifth Hospita
Record Dates: First submitted 2018-08-19; First posted 2018-09-07 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: NK Cell Mediated Immunity
MeSH Terms: interventions — Random Allocation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EGFR+NK+ (Experimental): The EGFR mutation positive patients were with the principles of randomized and NK cells treatment.
  Interventions: Biological: NK cells
- EGFR+NK- (No Intervention): The EGFR mutation positive patients were with the principles of randomized and without NK cells treatment .
- EGFR-NK+ (Experimental): The EGFR mutation negative patients were with the principles of randomized and NK cells treatment .
  Interventions: Biological: NK cells
- EGFR-NK- (No Intervention): The EGFR mutation negative patients were with the principles of randomized and without NK cells treatment.

INTERVENTIONS:
Biological: NK cells — NK cells were generated in good manufacturing practice (GMP) condition. In brief, PBMCs were isolated from 50mL patient's blood with Ficoll-Hypaque(Morecell Biomedical Co. Ltd., Shenzhen, China). Then the Human NK Cell Culture Kit (Cat. No.
  MCF-004, Morecell Biomedical Co. Ltd., Shenzhen, China) and Serum-free Medium for NK Cells (MCM-002, Morecell Biomedical Co. Ltd., Shenzhen, China) was used for induction of NK cells according to the manufacturer's instructions. Three days before NK cell transfusion, the NK cells were sampled and sent to detect the NK cell quality.
  Other Names: randomized
  Arms: EGFR+NK+; EGFR-NK+

SUMMARY:
This study was attempted to investigate the efficiency of NK cells immunotherapy on non-small cell lung cancer with and without EGFR mutation, and evaluated response rate (RR) and the progression-free survival (PFS).

DETAILED DESCRIPTION:
Investigators will enrolle 100 patients who met the enrollment criteria. 50 patients were clinically confirmed EGFR mutation positive. They were divided into two groups (group A and group C according to if accepted NK therapy) in accordance with the principles of randomized. The rest 50 patients which were EGFR mutation negative were also divided into two groups (group B and group D) in accordance with the principles of randomized to be paired respectively with group A and group C. Comparison of lymphocyte number, serum tumor related biomarkers, circulating Tumor Cell (CTC), KPS and survival curves was carried out before after NK cell immunotherapy. The safety and short-term effects were evaluated followed by the median PDA, response rate assessment.

ELIGIBILITY:
Inclusion Criteria:

The criteriaof the enrollment are as following: (1) expected survival>6 months; (2) age between35-75 years old; (3) KPS >45; (4) platelets>80 × 109/L, WBC>3 × 109/L, hemoglobin>90g/L, prothrombin time-international normalized ratio (0.8-1.5), adequate hepatic function (bilirubin < 20 μM, aminotransferase<60 U/L) and renal function (serum creatinine < 130 μM, serum urea <10 mM); (5) All patients confirmed by pathology and/or imaging;

Exclusion Criteria:

The absence of level 3 hypertension, severe coronary disease, myelosuppression, respiratory disease, acute or chronic infection, and autoimmune diseases. -

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Calculated the sum area of all tumors 3 months after NK treatment
  Based on the Response Evaluation Criteria Solid Tumors (RECIST), the therapeutic effect was divided into complete response (CR), partial response (PR),stable disease (SD), progressive disease (PD). Investigators calculated the sum area of all tumors 3 months after NK treatment. The recent curative effect must have been maintainedat >4 weeks; CR + PR denoted the effective response rate (RR).

SECONDARY OUTCOMES:
Detection of immune function | Before and 3 months after NK cell therapy
  Patients were detected Lymphocyte subgroups of 1ml peripheral blood by Flow cytometer (BD FACSCalibur), which inclunde the T cell number, CD4T cell number, CD8 T cell number and NK cell number.
Analysis of tumor biomarker CEA and CA125 levels in serum | Before and 3 months after NK cell therapy
  Patients were detected the Serum Carcinoembryonic antigen (CEA) and CA125 level by Elisa kit.Investigators compared the level of CEA and CA125 in serum before and 3 months after NK cell therapy to perform the therapeutic evaluation.
  factor to identify patients tumor recurrence.We then compared the level of CEA and CA125 in serum before and 3 months after NK cell therapy to perform the therapeutic evaluation.

OTHER OUTCOMES:
The endpoints of interest were progression-free survival (PFS). | The KPS scores were collected pre-treatment and at 12 months post-treatment.
  Investigators evaluated the Karnofsky Performance Status (KPS) according to the comprehensive assessment of clinical activity, disease level, and self-care ability.
  Status (KPS) according to the comprehensive assessment of clinical activity, disease level, and self-care ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Luohu Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes